CLINICAL TRIAL: NCT06610084
Title: The Effect of Hypno-breastfeeding and Progressive Muscle Relaxation Exercise on Breastfeeding Motivation and Breastfeeding Self-Efficacy in Primiparous Women Delivered by Caesarean Section
Brief Title: The Effect of Hypno Breastfeedıng and Progressıve Muscle Relaxatıon Exercıse on Breastfeedıng Self-Effıcacy and Breastfeedıng Motıvatıon
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: received comprehensive hypno-breastfeeding training
Sponsor: Tuğba Konukoğlu (Other)
Responsible Party: Sponsor-Investigator, Tuğba Konukoğlu, research assistant, Sanko University
Organization: Sanko University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SankoU-Nursing-TKY-01
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Breastfeeding Education
Keywords: breastfeeding; self efficacy; breastfeeding motivation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: This research is a randomised controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypno-breastfeeding (Experimental): The research was conducted in a total of 6 sessions. Session 1 (32nd week): After the introduction, hypno-breastfeeding practice was performed face-to-face.
  Session 2 (33rd-34th week): Hypno-breastfeeding practice was repeated with online interviews.
  Session 3 (35th week): Hypno-breastfeeding practice was repeated face-to-face. Session 4 (36th week): Hypno-breastfeeding practice was repeated online. Session 5 (37th week): Hypno-breastfeeding practice was repeated face-to-face. Session 6 (38th-40th week): Hypno-breastfeeding practice was performed in the ward at the 8th hour postpartum.
  Postpartum 2nd to 4th week: The audio recording prepared by the researcher was used for the hypno-breastfeeding application given to the mother. The researcher guided the mother to perform the application once a day and followed up with daily telephone calls.
  Translated with DeepL.com (free version)
  Interventions: Other: Hypno-breastfeeding
- progressive muscle relaxation exercise (Experimental): Applications for experimental group 2 (progressive muscle relaxation exercise) The research was conducted in a total of 6 sessions. Session 1 (32nd week): After the introduction, progressive muscle relaxation exercise was performed face-to-face.
  Session 2 (Week 33-34): Progressive muscle relaxation exercise was repeated with online interview.
  Session 3 Week 35: In Phase 3, the progressive muscle relaxation exercise was repeated face-to-face.
  Session 4 Week 36: Progressive muscle relaxation exercise was repeated online. Session 5 Week 37: Progressive muscle relaxation exercise, repeated face-to-face.
  Session 6 38.-40th Week: It was performed in the ward at the 8th hour postpartum.
  Postpartum 2nd to 4th week: The video prepared by the researcher was used for the progressive relaxation exercise training given to the mother. The researcher guided the mothers to perform the practice once a day and follow-up was ensured through daily telephone calls.
  Interventions: Other: progressive muscle relaxation exercise)

INTERVENTIONS:
Other: progressive muscle relaxation exercise) — Applications for experimental group 2 (progressive muscle relaxation exercise) The research was conducted in a total of 6 sessions. Session 1 (32nd week): After the introduction, progressive muscle relaxation exercise was performed face-to-face.
  Session 2 (Week 33-34): Progressive muscle relaxation exercise was repeated with online interview.
  Session 3 Week 35: In Phase 3, the progressive muscle relaxation exercise was repeated face-to-face.
  Session 4 Week 36: Progressive muscle relaxation exercise was repeated online. Session 5 Week 37: Progressive muscle relaxation exercise, repeated face-to-face.
  Session 6 38.-40th Week: It was performed in the ward at the 8th hour postpartum.
  Postpartum 2nd to 4th week: The video prepared by the researcher was used for the progressive relaxation exercise training given to the mother. The researcher guided the mothers to perform the practice once a day and follow-up was ensured through daily telephone calls.
  Arms: progressive muscle relaxation exercise
Other: Hypno-breastfeeding — Practices for experimental group 1 (Hypno-breastfeeding) The research was conducted in a total of 6 sessions. Session 1 (32nd week): After the introduction, hypno-breastfeeding practice was performed face-to-face.
  Session 2 (33rd-34th week): Hypno-breastfeeding practice was repeated with online interviews.
  Session 3 (35th week): Hypno-breastfeeding practice was repeated face-to-face. Session 4 (36th week): Hypno-breastfeeding practice was repeated online. Session 5 (37th week): Hypno-breastfeeding practice was repeated face-to-face. Session 6 (38th-40th week): Hypno-breastfeeding practice was performed in the ward at the 8th hour postpartum.
  Postpartum 2nd to 4th week: The audio recording prepared by the researcher was used for the hypno-breastfeeding application given to the mother. The researcher guided the mother to perform the application once a day and followed up with daily telephone calls.
  Arms: Hypno-breastfeeding

SUMMARY:
Topic: The World Health Organisation (WHO) states that breastfeeding is of great importance for the healthy growth and development of infants as well as for maternal health. Breast milk is a unique and irreplaceable food. Breast milk is the most natural food for infant nutrition and contains all the nutrients, vitamins and minerals needed by the baby. Breast milk provides sensory and cognitive development and helps to protect the baby against all kinds of infectious and chronic diseases . The benefits of breastfeeding are not limited to infant health. Breastfeeding is also of great importance for maternal and public health. According to TDHS 2018 data, the proportion of exclusively breastfed infants decreases rapidly with age, from 59% among 0-1 month-olds to 45% among 2-3 month-olds and 14% among 4-5 month-olds. Accordingly, it is observed that the rate of breastfeeding maintenance is low in Turkey.

Breastfeeding motivation and breastfeeding self-efficacy are modifiable factors in initiating and maintaining breastfeeding. It has been found that breastfeeding duration of mothers with high breastfeeding motivation is longer.. In studies, breastfeeding self-efficacy of adult women has been defined as an important variable affecting breastfeeding outcomes. Especially prenatal breastfeeding self-efficacy has been shown to predict breastfeeding intentions and the predicted length of breastfeeding. In the literature, it was reported that mothers with low breastfeeding self-efficacy perception discontinued breastfeeding in a short period of time after delivery, whereas mothers with high breastfeeding self-efficacy perception did not have any difficulty in initiating and maintaining breastfeeding.

Pharmacological and nonpharmacological interventions have been focused on to increase prolactin secretion and breast milk production of mothers in the postpartum period.These interventions will decrease the stress and anxiety of the mother and help breastfeeding by increasing breastfeeding motivation and breastfeeding self-efficacy. Therefore, nonpharmacological methods for increasing lactation and elimination of breast problems are important in terms of both breastfeeding and continuity of breastfeeding. Practices used to increase lactation include kangaroo care, back massage, yoga, breast massage, compression, acupuncture, acupressure, music therapy, aromatherapy, herbal tea use and galactagogues techniques. Hypno-breastfeeding and progressive muscle relaxation exercise used in this study are among these practices. Hypno-breastfeeding is hypnosis that helps to increase breast milk and is performed with a hypnotherapist who pays attention to the unity of body, mind and spirit and its philosophy is based on hypnosis and breastfeeding programme.Progressive muscle relaxation exercise has also been found to increase breastfeeding self-efficacy. As a result of active contraction and passive relaxation of 16 muscle groups, the person relaxes physiologically by decreasing the activity of the sympathetic nervous system and increasing the activity of the parasympathetic nervous system. 16 muscle groups actively contracted and passively relaxed, it was found that the person relaxed physiologically by decreasing the activity of the sympathetic nervous system and increasing the activity of the parasympathetic nervous system. Relaxation has been shown to effectively improve perceived stress levels and to be effective in helping people control their emotions and behaviours in many situations such as pain, labour, anxiety and insomnia. With the comfort provided by relaxation, the mother's orientation towards breastfeeding will increase. Hypno-breastfeeding and progressive muscle relaxation exercise will have an effect on increasing breastfeeding motivation and breastfeeding self-efficacy.

DETAILED DESCRIPTION:
This research is a randomized controlled experimental study. The research will be conducted in SANKO University Sani Konukoğlu Application and Research Hospital NST unit and Gynecology Service in Gaziantep. The population of the study will consist of pregnant women admitted to SANKO University Sani Konukoğlu Practice and Research Hospital Obstetrics Outpatient Clinic. When power analysis was performed, the minimum sample size per group was found to be 16. It is planned to take a minimum of 40 people per group. Data Collection Tools "Personal Information Form", 'Prenatal Breastfeeding Self-Efficacy Scale', 'Primiparous Breastfeeding Motivation Scale' and 'Breastfeeding Self-Efficacy Scale Short Form' were used to collect the data.

Personal Information Form This form prepared by the researcher consists of a total of 20 questions that can determine the socio-demographic and obstetric characteristics of pregnant women.

Prenatal Breastfeeding Self-Efficacy Scale It was developed by Wells et al. in 2006 to determine pregnant women's perceptions of breastfeeding self-efficacy. It was adapted into Turkish by Aydın and Pasinlioğlu in 2016. The scale consists of a total of 20 items and has no sub-dimensions. The scale is 5-point Likert type. The items of the scale are; "Not at all sure" (1 point), "Somewhat sure" (2 points), "Quite sure" (3 points), "Very sure" (4 points), "Completely sure" (5 points). There are no reverse scored items in the scale. The lowest score that can be obtained from the scale is 20 and the highest score is 100. The scale has no cut-off point. An increase in the score obtained from the scale indicates an increase in the perception of breastfeeding self-efficacy. The Cronbach's alpha coefficient of the Turkish version of the scale is 0.86. The Cronbach's Alpha coefficient in this study was 0.95 Primiparous Breastfeeding Motivation Scale It was developed by Stockdale et al. in 2013 to determine the factors affecting breastfeeding motivation in primiparous women. The scale was adapted into Turkish by Akçay and Demirgöz Bal in 2019. The scale consists of a total of 29 items and is 7-point Likert-type. The scale has 4 sub-dimensions.

Breastfeeding Self-Efficacy Scale Short Form It is a 33-item scale prepared by Dennis and Faux (127) in 1999 to assess breastfeeding self-efficacy levels. A short form of the 14-item Breastfeeding Self-Efficacy Scale was developed by Aluş-Tokat et al. in 2010. The scale is a 5-point Likert scale. The lowest score that can be obtained from the scale is 14 and the highest score is 70. The scale has no cut-off point. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy. The Cronbach Alpha value of the scale is 0.94.

Implementation of the Study: The data will be collected face-to-face by the researcher herself. Patients who meet the inclusion criteria will be included in the control and intervention groups using face-to-face interview method. The implementation of the study will take place in 7 stages for 2 intervention groups (Hypno-breastfeeding and progressive muscle relaxation exercise).

Pregnant women in the experimental and control groups will receive routine breastfeeding education during pregnancy follow-up. After cesarean delivery, pregnant women will receive routine postpartum nursing care and the interventions, medication/order list, time and method of administration will be applied in a standardized manner. Pregnant women in the control group will not receive any intervention. The interventions applied to the experimental groups are given below. Before the interventions were implemented, the prepared materials were sent to the experts via e-mail and expert opinion was obtained. For hypno-breastfeeding; training chart, relaxation text and audio recording, for progressive muscle relaxation exercise, training chart, relaxation text and video were prepared. Necessary corrections were made in the relaxation texts and schedules in line with expert opinions. Hypno-breastfeeding and progressive muscle relaxation exercise practices will be performed by the researcher herself.

Evaluation of the Data IBM SPSS Statistics 22 package program will be used for data analysis. In statistical evaluation; categorical measurements will be summarized as number and percentage, continuous measurements will be summarized as mean, deviation and minimum-maximum. Chi-square test and Fischer's Exactness Test will be used for comparisons of categorical variables. The conformity of the variables to the normal distribution will be examined using visual (histograms and probability graphs) and analytical methods (Kolmogorov-Smirnov/Shapiro-Wilk Tests). One-way Anova test will be used for more than two variables in groups that conform to normal distribution, while Kruskall Wallis tests will be used for more than two variables in groups that do not conform to normal distribution. Bonferroni analysis will be used in Post Hoc analyzes to determine the source of the difference between groups. The results will be evaluated at 95% confidence interval and p<0.05 error level.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Literate,
* Can understand and speak Turkish,
* A singular pregnancy,
* Gestation period of 32 weeks or more,
* She's scheduled to give birth by caesarean section,
* Volunteered to participate in the research, primiparous pregnant women were included in the study.

Exclusion Criteria:

* - Having developed any complications in herself and the newborn during pregnancy, labour and postnatal period,
* Chronic opioid, antidepressant, psychoactive drug users,
* Communication problems primiparous pregnant women were not included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study was planned on pregnant women
Enrollment: 120 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale Short Form | 3 month
  It is a 33-item scale prepared by Dennis and Faux (127) in 1999 to assess breastfeeding self-efficacy levels. A short form of the 14-item Breastfeeding Self-Efficacy Scale was developed by Aluş-Tokat et al. in 2010. The scale is 5-point Likert type. The lowest score that can be obtained from the scale is 14 and the highest score is 70. The scale has no cut-off point. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy. Cronbach Alpha value of the scale is 0.94. (Aluş-Tokat & Okumuş, 2010).

SECONDARY OUTCOMES:
Breastfeeding Self-Efficacy Scale | 3 month
  Prenatal Breastfeeding Self-Efficacy Scale It was developed by Wells et al. in 2006 to determine the breastfeeding self-efficacy perceptions of pregnant women. It was adapted into Turkish by Aydın and Pasinlioğlu in 2016. The scale consists of a total of 20 items and has no sub-dimensions. The scale is 5-point Likert type. The items of the scale are; 'I am not sure at all' (1 point), 'I am a little sure' (2 points), 'I am quite sure' (3 points), 'I am very sure' (4 points), 'I am completely sure' (5 points). There are no reverse scored items in the scale. The lowest score that can be obtained from the scale is 20 and the highest score is 100. The scale has no cut-off point. An increase in the score obtained from the scale indicates an increase in the perception of breastfeeding self-efficacy. The Cronbach's alpha coefficient of the Turkish version of the scale is 0.86. The Cronbach's Alpha coefficient in this study was 0.95.
Primiparous Breastfeeding Motivation Scale | 3 month
  Primiparous Breastfeeding Motivation Scale It was developed by Stockdale et al. in 2013 to determine the factors affecting breastfeeding motivation in primiparous women. The scale was adapted into Turkish by Akçay and Demirgöz Bal in 2019. The scale, which consists of a total of 29 items, is 7-point Likert type. The scale has 4 sub-dimensions

CONTACTS AND LOCATIONS:
Locations (1):
- SANKO Unıversity, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study ProtocolStatistical Analysis Plan (SAP)
  Informed Consent Form (ICF)
  Clinical Study Report (CSR)
  Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: June 24-March 28
Access Criteria: ipd other researcher will access the full research protocol by email from the researcher.